CLINICAL TRIAL: NCT00628290
Title: Evaluation of the Antipsychotic Efficacy of the Phytocannabinoid Cannabidiol in Treating Acute Schizophrenic Psychosis. A Double-Blind, Controlled Clinical Trial
Brief Title: Evaluation of the Antipsychotic Efficacy of Cannabidiol in Acute Schizophrenic Psychosis
Acronym: CBD-CT1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Cologne (Other)
Responsible Party: Dr. F. Markus Leweke, University of Cologne
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CBD-CT1; SMRI Grant ID: 00-093
Record Dates: First submitted 2008-02-26; First posted 2008-03-05 (Estimated); Last update posted 2008-03-18 (Estimated); Status verified 2008-01

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Cannabidiol; Amisulpride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Cannabidiol
- 2 (Active Comparator)
  Interventions: Drug: Amisulpride

INTERVENTIONS:
Drug: Cannabidiol — Capsules, 3 times daily, 200 mg, 4 weeks
  Arms: 1
Drug: Amisulpride — Capsules, 3 times daily, 200 mg, 4 weeks
  Arms: 2

SUMMARY:
A controlled, randomized study on the treatment of schizophrenic psychosis with cannabidiol, a phytocannabinoid is performed. This approach is based upon recent findings indicating that the human endogenous cannabinoid system is significantly involved in the pathogenesis of schizophrenia. Our group has shown, for example, that Δ9-tetrahydrocannabinol (Δ9-THC) is able to provoke schizophrenia-like psychotic symptoms in healthy volunteers. This, as well as the capability of Δ9-THC to exacerbate productive psychotic symptoms in schizophrenic patients, has recently been confirmed by others. Furthermore, we found that the en-dogenous brain constituent anandamide, an endogenous Δ9-THC agonist, is significantly elevated in the CSF of schizophrenic patients. Cannabinergic substances such as anandamide may enhance dopaminergic neurotrans-mission by increasing dopamine turnover. They may also influence the onset or course of schizophrenia by as yet unidentified mechanisms We seek to investigate the efficacy of cannabidiol in the treatment of schizophrenic and schizophreniform psy-choses, because there is evidence that CB1 antagonists such as SR141716 and cannabidiol have antipsychotic effects comparable to those of classic neuroleptic drugs. Furthermore, cannabidiol is well tolerated showing few side effects in humans. Cannabidiol may serve as an antipsychotic medication that is not primarily based upon an antidopaminergic but upon different mechanisms, especially anticannabinergic ones. It may therefore be an effec-tive medication in at least a subgroup of schizophrenic and schizophreniform patients and may be expected to show additional anxiolytic effects and only minor side effects.

The control condition in this parallel design will be an established neuroleptic treatment with amisulpride that is primarely an antidopaminergic drug. Thus, we will study not only the antipsychotic efficacy of cannabidiol, but we will also compare the effects of both treatment strategies on side effects and neuropsychological functioning.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of schizophrenia or schizophreniform psychosis according to DSM-IV.
* BPRS score >36 and BPRS psychosis cluster > 12.
* Ability to provide written informed consent.
* Participants are required an adequate contraception.

Exclusion Criteria:

* Any severe neurological or somatic disorder.
* Other psychiatric disorders including addictive disorders.
* Positive urine drug screening for any compound except benzodiazepines.
* No pregnancy or breast feeding.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2002-10; Primary Completion 2004-11 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Change in BPRS total value. | 4 weeks

SECONDARY OUTCOMES:
Change in PANSS scores. | 4 weeks
EPS | 4 weeks
Weight gain | 4 weeks
Prolactin levels in serum | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Franz-Markus Leweke, MD, Principal Investigator — University of Cologne, Dept. of Psychiatry and Psychotherapy
Locations (1):
- University of Cologne, Dept. of Psychiatry and Psychotherapy, Cologne, North Rhine-Westphalia, Germany

REFERENCES:
- [Derived] Leweke FM, Rohleder C, Gerth CW, Hellmich M, Pukrop R, Koethe D. Cannabidiol and Amisulpride Improve Cognition in Acute Schizophrenia in an Explorative, Double-Blind, Active-Controlled, Randomized Clinical Trial. Front Pharmacol. 2021 Apr 29;12:614811. doi: 10.3389/fphar.2021.614811. eCollection 2021. PMID 33995015
- See also: Related Info — http://www.ecnp.net